CLINICAL TRIAL: NCT06610006
Title: Combined Effects of Isometric Wall Squats and High Intensity Interval Training on Rate Pressure Product in Normotensive and Pre-hypertensive Sedentary Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/34
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pre Hypertension
MeSH Terms: conditions — Prehypertension | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group(interventional group) will be doing High Intensity Training (HIIT) and Isometric Wall Squat and the other group (control group) will be doing High intensity Interval Training (HIIT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Interval Training (Active Comparator): Participants will begin with warm-up exercises for 5-7 mins before the session. Then they will begin high intensity interval training on treadmill with moderate intensity (40-60%HRR) in week 1 to achieve the baseline fitness level and from week 2 to 5 they will progress to high intensity with setting the lower target HR 40-60%HRR and upper target HR 80-85%HRR with 1:4 work to rest ratio followed by 5-7 min of cool-down period.A total of 15 sessions for thrice a week on alternative days for 5 consecutive weeks will be given
  Interventions: Procedure: High Intensity Interval Training (HIIT)
- High Intensity Interval Training (HIIT) and Isometric Wall Squat (Experimental): High intensity interval training on treadmill with moderate intensity (40-60%HRR) in week 1 to achieve the baseline fitness level and from week 2 to 5 they will progress to high intensity with setting the lower target HR 40-60%HRR and upper target HR 80-85%HRR with 1:4 work to rest ratio. For isometric wall squat, each training session will be composed of 4 × 2-min bouts of IWS followed by 2-min rest periods At the end of each bout, participants will be given an RPE score. This score will then be compared to a target RPE value and zone for each bout, There will be total 15 sessions thrice a week for 5 weeks.
  Interventions: Procedure: High Intensity Interval Training (HIIT); Procedure: Isometric Wall Squat

INTERVENTIONS:
Procedure: High Intensity Interval Training (HIIT) — High intensity interval training on treadmill with moderate intensity (40-60%HRR) in week 1 to achieve the baseline fitness level and from week 2 to 5 they will progress to high intensity with setting the lower target HR 40-60%HRR and upper target HR 80-85%HRR with 1:4 work to rest ratio followed by 5-7 min of cool-down period..A total of 15 sessions of high intensity interval training alone , for thrice a week on alternative days for 5 consecutive weeks will be given. Warm-up session consisting of stretching exercises prior to intervention and cool down session after intervention will also be done and vitals before and after the session will be taken.
Procedure: Isometric Wall Squat — For isometric wall squat, each training session will be composed of 4 × 2-min bouts of IWS followed by 2-min rest periods. In first week, participants will do squat training or there will be a protocol for selecting exercise intensity in which participants will be given 30-s to perform a wall squat to select a position that they predict would elicit an target RPE score by varying the squat height. Based on the final squat height and RPE score, after bout 4, participants will be given a starting squat height for training session 1 and will then be progressed in each week
  Arms: High Intensity Interval Training (HIIT) and Isometric Wall Squat

SUMMARY:
Hypertension is leading yet preventable risk factor for cardiovascular disease and all-cause mortality worldwide. Prehypertension identifies those at high risk of developing HTN, prompting intervention to prevent or delay the onset of the disease. High intensity interval training (HIIT) is a time efficient mode of training with established benefits, while Isometric wall squats (IWS) also provide a range of proven benefits and advantages, but their combined effect on BP measures is yet to be determined.Hence the objective of this study is to compare the effects of isometric wall squats along with high intensity interval training versus high intensity interval training alone on rate pressure product, SBP and DBP, heart rate and anthropometric measures in normotensive and pre-hypertensive sedentary adults

DETAILED DESCRIPTION:
Pre-Hypertension is not a disease itself rather it categorizes those who are at the risk of developing hypertension in future. By targeting pre-hypertensive and normotensive individuals we are focusing on preventive measures, potentially reducing incidence of HTN and cardiovascular conditions in future. If found effective, this study can help in providing training protocols while also decreasing the risk of hypertension in future.A total of 15 sessions of high intensity interval training alone in one group and combination of high intensity interval and isometric wall squat in other group, for thrice a week on alternative days for 5 consecutive weeks will be given.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female adults aged 18-45 years.
* Participants lying in Low PA (inactive) category on basis of IPAQ.
* Pre-hypertensive adults:
* SBP- 120 mmHg or more and <140 mmHg
* DBP of 80 mmHg or more and < 90 mmHg.
* Normotensive adults: SBP < 120 mmHg and DBP < 80 mmHg. Exclusion Criteria
* Diagnosed with any current infections.
* Subjects with any diagnosed cardiovascular or respiratory conditions.
* Subjects with diagnosed musculoskeletal or neurological conditions which hinder participation in physical activity program.
* Active Smokers
* Those with any contraindication to exercise testing or training.
* Pregnant females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate Pressure Product | 5 weeks
  Measured by multiplying Heart Rate and Systolic Blood Pressure
Blood Pressure(SBP and DBP) | 5 weeks
  Evaluation will be done using sphygmomanometer
Heart rate | 5 weeks
  Heart Rate will be measured using pulse oximeter.
Anthropometric Measures Waist circumference | 5 weeks
  Measuring Tape will be used to measure Waist circumference
Anthropometric Measures hip circumference | 5 weeks
  Measuring Tape will be used to measure hip circumference
Anthropometric Measures Waist to hip ratio | 5 weeks
  Ratio of waist circumference and hip circumference
BMI | 5 weeks
  Body mass index ratio of weight and height

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan